CLINICAL TRIAL: NCT04754646
Title: A Randomized, Controlled, Single-blinded, Within-subject (Split-face), Multicenter, Prospective Clinical Study to Evaluate the Effectiveness and Safety of Using the Dermal Filler RHA®4 Injected With a Cannula or With a Sharp Needle for the Treatment of Moderate to Severe Nasolabial Folds
Brief Title: RHA® 4 NLF Cannula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEO-RHA-2001
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Wrinkle; Nasolabial Fold; Aging
Keywords: Dermal Filler; Hyaluronic acid; Cannula; Nasolabial folds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded-Live Evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- RHA®4 - Cannula (Experimental)
  Interventions: Device: Split-face injection of RHA® 4 with a cannula into a single NLF.
- RHA®4 - Needle (Active Comparator)
  Interventions: Device: Split-face injection of RHA® 4 with a needle (TSK 27G x ½") into the contralateral NLF.

INTERVENTIONS:
Device: Split-face injection of RHA® 4 with a cannula into a single NLF. — RHA® 4 is a sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus equi bacteria, formulated to a concentration of 23 mg/mL and 0.3% w/w lidocaine in a physiologic buffer.
  Up to 3.0 mL injected per NLF (mid-dermis to deep-dermis). Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
  The brand of cannula used for injection is up to the discretion of the Treating Investigator (TI), providing the cannula is registered for use by the US FDA.
  Arms: RHA®4 - Cannula
Device: Split-face injection of RHA® 4 with a needle (TSK 27G x ½") into the contralateral NLF. — RHA® 4 is a sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus equi bacteria, formulated to a concentration of 23 mg/mL and 0.3% w/w lidocaine in a physiologic buffer.
  Up to 3.0 mL injected per NLF (mid-dermis to deep-dermis). Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
  Arms: RHA®4 - Needle

SUMMARY:
This is a randomized, controlled, single-blinded, within-subject (split-face), multicenter, prospective study to investigate whether RHA®4 injected in NLFs with a cannula is non-inferior to RHA®4 injected in NLFs with a sharp needle (27G x ½") for the correction of moderate to severe NLFs as determined by the Blinded Live Evaluator (BLE) using the Teoxyne NLF-WSRS (proprietary, validated NLF Wrinkle Severity Rating Scale) at 12 weeks from last treatment.

At Visit 1 (Week 0), RHA®4 injected with cannula will be administered in a random sequence (first or second injection) and side of the face (left or right NLF) and RHA®4 injected with a sharp needle will be administered to the other side. The TI will administer study devices and will be unblinded to treatment allocation. Blinded assessments of effectiveness will be conducted by the BLE (Blinded Live Evaluator).

4 weeks following initial treatment, subjects will attend Visit 2 and receive, if necessary, touch-up treatments (using a needle or cannula as per the subject's initial treatment assignment).

Subjects receiving touch-up treatments at Week 4 (Visit 2) will attend a new Visit 2b (4 weeks following touch-up treatment); subject not receiving touch-up treatment will not attend Visit 2b.

After each injection (initial treatment or touch-up), subjects will receive a safety follow-up call from the study site within 3-day.

Subjects will then attend scheduled in-office study visits at 8 (Visit 3) and 12 weeks (Visit 4) following last treatment (initial treatment or touch-up) where safety and effectiveness assessments will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, 22 years of age or older.
* Female subjects of childbearing potential must have a negative UPT and practice a reliable method of contraception throughout the study.
* Moderate to severe bilateral nasolabial folds (grade 3 or 4 on the five-point NLF-WSRS). BLE and TI must independently agree that the criterion is met; however, strict concordance of severity not required. BLE assessments will be used for the primary endpoint. If TI and BLE do not agree on eligibility, or if their assessments differ by ≥2 grades, the subject will not be eligible.
* Nasolabial folds of the same NLF-WSRS grade on the left and right sides of the face.
* Willing to abstain from facial aesthetic procedures/therapies that could interfere with the study evaluations.
* Able to follow study instructions and complete all required visits.
* Sign the IRB-approved ICF, Photographic Release Form, the Authorization for Use and release of Health and Research Study Information (HIPAA) form, and if applicable, the California Experimental Research Subject's Bill of Rights prior to any study-related procedures being performed.

Exclusion Criteria:

* Known hypersensitivity or previous allergic reaction to any component of the study devices.
* Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, or history of anaphylactic shock.
* History of active chronic debilitating systemic disease that, in the opinion of the investigator, would make the subject a poor candidate in the study.
* History of connective tissue disease.
* Malignancy (excluding non-melanoma skin cancer) within the past 5 years.
* History of skin cancer in the treatment area.
* Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
* Exposure to any other investigational drug/device within 90 days of entering the study or planning to participate in another investigation during the course of the study.
* Study staff or close relative to study staff (e.g., parents, children, siblings, or spouse)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - United States, California, Encinitas, California
  - United States, Florida, West Palm Beach, Florida
  - United States, North Carolina, Chapel Hill, North Carolina
  - United States, Tennessee, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Bilateral Treatment of RHA® 4 With a Cannula Vs RHA® 4 With a Needle: Split-face injection of RHA® 4 with a cannula into the NLF on one side of the face and RHA® 4 with a needle into the NLF on the opposide side of the face.
  RHA®4 injected with cannula was administered in a random sequence (first or second injection) and side of the face (left or right NLF) and RHA®4 injected with a sharp needle was administered to the other side.
  The brand of cannula used for injection is up to the discretion of the Treating Investigator (TI), providing the cannula is registered for use by the US FDA.
Period: Overall Study
Arm/Group | Bilateral Treatment of RHA® 4 With a Cannula Vs RHA® 4 With a Needle
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bilateral Treatment of RHA® 4 With a Cannula Vs RHA® 4 With a Needle
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 39
  More than one race | 0
  Unknown or Not Reported | 1
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type as determined by the Treating Investigator on the skin tone scale developed to classify skin coloring and response to ultraviolet (UV) radiation. The scale contains 6 grades:
  I: Pale white skin; Always burns, does not tan. II: Fair skin; Burns easily, tans poorly. III: Darker white skin; Tans after initial burn. IV: Light brown skin; Burns minimally, tans easily. V: Brown skin; Rarely burns, tans darkly easily. VI: Dark brown or black skin; Never burns, always tans darkly.
  Participants
    Fitzpatrick Skin Type I-III | 38
    Fitzpatrick Skin Type IV-VI | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in NLF-WSRS Score Between Baseline and Week 12 After Last Treatment as Assessed by the BLE
Description: Non-inferiority of RHA®4 injected with a cannula to the change from Baseline for subjects treated with RHA®4 injected with a needle at 12 weeks after last treatment (initial or touch-up; up to 16 weeks post-baseline)) as assessed by the BLE using the NLF-WSRS.
  NLF-WSRS (Nasolabial Folds - Wrinkle Severity Rating Scale) is a proprietary validated 5-grade scale with 1 being "Absent" and 5 being "Extreme".
  An NLF-WSRS change of >1 grade will be considered clinically significant.
Time Frame: Week 12 after last treatment
Population: Per Protocol population (Of the 50 subjects randomized, 4 subjects experienced at least one major protocol deviation that resulted in their exclusion from the PP population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 46 | 46
score on a scale | -1.61 (0.21) | -1.65 (0.21)

2. Secondary Outcome: Change in Score From Baseline in the Nasolabial Folds Severity Rated by the Treating Investigator (TI) at Weeks 4, 8 and 12 After Last Treatment Using the NLF-WSRS.
Description: NLF-WSRS (Nasolabial Folds - Wrinkle Severity Rating Scale) is a proprietary validated 5-grade scale with 1 being "Absent" and 5 being "Extreme".
Time Frame: Weeks 4, 8 and 12 after last treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
score on a scale
  Week 4 after last treatment | -1.2 (0.56) | -1.3 (0.59)
  Week 8 after last treatment | -1.5 (0.65) | -1.6 (0.70)
  Week 12 after last treatment | -1.5 (0.58) | -1.6 (0.67)

3. Secondary Outcome: Number of Responders (Change of ≥1-grade From Baseline in the Naso-labial Folds Severity) as Assessed by the Blinded Live Evaluator (BLE) at Week 12 After Last Treatment Using the NLF-WSRS.
Description: NLF-WSRS (Nasolabial Folds- Wrinkle Severity Rating Scale) is a proprietary validated 5-grade scale with 1 being "Absent" and 5 being "Extreme".
Time Frame: Week 12 after last treatment
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
Participants | 47 | 47

4. Secondary Outcome: Number of Responders (Change of ≥1-grade From Baseline in the Naso-labial Folds Severity) as Assessed by the Treating Investigator (TI) at Weeks 4, 8 and 12 After Last Treatment Using the NLF-WSRS.
Description: NLF-WSRS (Nasolabial Folds- Wrinkle Severity Rating Scale) is a validated 5-grade scale with 1 being "Absent" and 5 being "Extreme"
Time Frame: Weeks 4, 8 and 12 after last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
Participants
  Week 4 after last treatment | 47 | 48
  Week 8 after last treatment | 48 | 48
  Week 12 after last treatment | 49 | 49

5. Secondary Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the Blinded Live Evaluator (BLE) at 12 Weeks Following Last Treatment.
Description: The Global Aesthetic Improvement (GAI) is a subjective, balanced, 5-point dynamic scale assessing cosmetic improvement. Possible scores range from "much improved", "improved", "no change", "worse", to "much worse". The GAI will be assessed using the pre-injection baseline photograph. Each side of the face will be assessed independently.
Time Frame: Week 12 after last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
Participants | 50 | 50

6. Secondary Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the Treating Investigator (TI) at 4, 8 and 12 Weeks Following Last Treatment.
Description: as for outcome 5
Time Frame: Weeks 4, 8 and 12 after last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
Participants
  Week 4 after last treatment | 46 | 47
  Week 8 after last treatment | 50 | 50
  Week 12 after last treatment | 49 | 47

7. Secondary Outcome: Number of Subjects Who Scored Themselves Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale at 4, 8 and 12 Weeks Following Last Treatment.
Description: The Global Aesthetic Improvement (GAI) is a subjective, balanced, 5-point dynamic scale assessing cosmetic improvement. Possible scores range from "much improved", "improved", "no change", "worse", to "much worse". The GAI will be assessed using the pre-injection baseline photograph. Each side of the face was assessed independently.
  Subjects will be instructed: "Use a mirror to compare your face to the photograph provided to you and rate the degree of aesthetic improvement by using the following scale".
Time Frame: Weeks 4, 8 and 12 after last treatment
Population: ITT Population: 50 subjects
  1 missing data at week 4
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
Participants
  Week 4 after last treatment: number analyzed (Participants) | 49 | 49
  Week 4 after last treatment | 46 | 47
  Week 8 after last treatment | 48 | 47
  Week 12 after last treatment | 47 | 48

8. Secondary Outcome: Number of Subjects "Satisfied" or "Very Satisfied" With Study Treatment Using the Subject Satisfaction Scale at 4, 8 and 12 Weeks Following Last Treatment.
Description: The Subject Satisfaction Scale is a subjective, balanced, 5-point scale assessing subject satisfaction with study treatment. Possible scores range from with 1 (very satisfied) to 5 (very dissatisfied).
Time Frame: Weeks 4, 8 and 12 after last treatment
Population: ITT Population: 50 subjects
  1 missing data at week 4
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
Participants
  Week 4 after last treatment: number analyzed (Participants) | 49 | 49
  Week 4 after last treatment | 46 | 45
  Week 8 after last treatment | 48 | 48
  Week 12 after last treatment | 45 | 48

9. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the FACE-Q | Aesthetics© (Nasolabial Folds Domain) Questionnaire. The FACE-Q Measures the Experience and Outcomes of Aesthetic Facial Procedures From the Patient's Perspective.
Description: The FACE-Q | Aesthetics© questionnaire is composed of 5 questions with a score linked to answers (1 being 'Not at all' and 4 being 'Extremely').
  The subject will be instructed as follows: "These questions ask about how you look right now. For each question, circle only one answer. With your nasolabial folds in mind (the deep lines that run downward from the sides of your nose), in the past week, how much have you been bothered by:", and will provide response.
  To calculate the FACE-Q, outcomes from all 5 questions were pooled, data were transformed so that higher scores reflected a superior (positive) outcome, and adapted to a scale of 100 units (i.e. worst/lowest score = 0, best/highest score = 100).
Time Frame: Weeks 4, 8 and 12 after last treatment
Population: ITT Population: 50 subjects
  1 missing data at week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
score on a scale
  Week 4 after last treatment: number analyzed (Participants) | 49 | 49
  Week 4 after last treatment | 35.8 (28.17) | 37.8 (26.71)
  Week 8 after last treatment | 40.0 (27.52) | 42.0 (27.29)
  Week 12 after last treatment | 40.7 (25.61) | 42.3 (27.93)

10. Secondary Outcome: Number of Participants Receiving Initial and Touch-Up Treatment Sessions to Obtain an Optimal Cosmetic Results as Judged by the Treating Investigator
Description: Number of subjects receiving treatment (initial and touch up)
Time Frame: Baseline (Week 0, Visit 1) and Touch-up (Week 4, Visit 2)
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
Participants
  Baseline (initial treatment) | 50 | 50
  Touch up (week 4) | 20 | 17

11. Secondary Outcome: Total Volume Per NLF to Obtain an Optimal Cosmetic Results as Judged by the Treating Investigator.
Time Frame: Baseline (Week 0) and Touch-up (Week 4)
Population: ITT: 50 subjects 20 subjects received a touch-up injection with cannula 17 subjects recieved a touch-up injection with needle
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
mL
  Baseline (Week 0) | 1.37 (0.48) | 1.40 (0.45)
  Touch Up (Week 4): number analyzed (Participants) | 20 | 17
  Touch Up (Week 4) | 0.85 (0.38) | 0.78 (0.41)
  Total | 1.71 (0.64) | 1.67 (0.63)

12. Secondary Outcome: NLF Symmetry as Assessed by the Blinded-live Evaluator at Baseline and 12 Weeks Following Last Treatment.
Description: NLF symmetry will be assessed for right and left NLF by answering the question "Are the NLFs symmetric or asymmetric?" (answer = symmetric or asymmetric answer). If asymmetric, the asymmetry will be further assessed as mild, moderate or severe.
Time Frame: Baseline (Week 0) and Week 12 after last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Treatment of RHA® 4 With a Cannula Vs RHA® 4 With a Needle
Number analyzed (Participants) | 50
Participants
  Symmetric at Baseline (post treatment) | 50
  Symmetric at Week 12 after last treatment | 47

13. Secondary Outcome: NLF Symmetry as Assessed by the Treating Investigator at Baseline 4, 8 and 12 Weeks Following Last Treatment.
Description: NLF symmetry will be assessed by the TI for right and left NLF by answering the question "Are the NLFs symmetric or asymmetric?" (answer = symmetric or asymmetric answer). If asymmetric, the asymmetry will be further assessed as mild, moderate or severe.
Time Frame: Weeks 4, 8 and 12 after last treatment
Population: ITT population: 50 subjects
  1 missing value at week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Treatment of RHA® 4 With a Cannula Vs RHA® 4 With a Needle
Number analyzed (Participants) | 50
Participants
  Symmetric at baseline (post treatment) | 50
  Symmetric at Week 4 after last treatment: number analyzed (Participants) | 49
  Symmetric at Week 4 after last treatment | 33
  Symmetric at Week 8 after last treatment | 40
  Symmetric at Week 12 after last treatment | 38

14. Secondary Outcome: NLF Symmetry as Assessed by the Subject at Baseline, 4, 8 and 12 Weeks Following Last Treatment.
Description: as for outcome 12
Time Frame: Weeks 4, 8 and 12 after last treatment
Population: ITT popualtion : 50 subjects
  1 missing value at week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Treatment of RHA® 4 With a Cannula Vs RHA® 4 With a Needle
Number analyzed (Participants) | 50
Participants
  Symmetric at Baseline (post treatment) | 41
  Symmetric at Week 4 after last treatment: number analyzed (Participants) | 49
  Symmetric at Week 4 after last treatment | 25
  Symmetric at Week 8 after last treatment | 32
  Symmetric at Week 12 after last treatment | 31

15. Secondary Outcome: Number of Participants With Adverse Events (AEs) for the Safety Evaluation of RHA® 4
Description: The Treating Investigator will assess adverse events and record details of seriousness, severity, duration, and action taken with the study device, and relationship to the study device. AEs will be reported from the time of consent until week 12 of the last treatment.
  An AE is any untoward medical occurrence in a subject administered the study device and which may, but does not necessarily, have a causal relationship with the device. An AE can therefore be any unfavorable or unintended sign (for example an abnormal laboratory finding), symptom or disease temporally associated with the use the study device, whether or not considered related to that device.
Time Frame: Baseline through Week 12 after last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
Participants
  Any Treatment Emergent Adverse Event | 27 | 33
  Any Treatment Related Adverse Event | 23 | 29
  Any Serious Adverse Event | 0 | 0
  Any Treatment Related Serious Adverse Event | 0 | 0
  Any Unexpected Adverse Device Effects | 0 | 0
  Any Adverse Effects of Special Interest | 3 | 3

16. Secondary Outcome: Number of Post-Injection Treatment Responses (From Common Treatment Responses (CTR) Diary) for the Safety Evaluation of RHA® 4.
Description: The subjects will receive a diary booklet and instructions for recording his/her observations of the Common Treatment Responses of the study treatments for the first 28 days after treatment. The diary will be discussed during telephone follow-up visit. Subjects should complete the diary at approximately the same time each day (i.e., am or pm).
  The subject diary captures the following Common Treatment Responses (CTR) that occur following the injection of a dermal filler; specifically, redness, pain, tenderness, firmness, swelling, lumps/bumps, bruising, itching, discoloration, and "other".
  The 28-day patient CTR diary includes a detailed glossary describing all signs/symptoms listed in the diary; an option was provided to rate "other" if the subject experienced a sign/symptom that is not listed.
  The table presents the number of subjects experiencing at least 1 Common Treatment Response (CTR).
Time Frame: During 28 days after initial treatment and touch-up, so a total of 42 days post-baseline if the subject received a touch-up
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
Participants
  Bruising | 10 | 27
  Discoloration | 9 | 16
  Firmness | 40 | 43
  Itching | 10 | 17
  Lumps/Bumps | 33 | 45
  Pain | 21 | 30
  Redness | 21 | 33
  Swelling | 36 | 41
  Tenderness | 38 | 44

17. Secondary Outcome: Assessment at Each Injection Visit (Initial Inejction and Touch-up) of Injection Site Pain Felt by the Patient for the Safety Evaluation of RHA® 4 Immediately After Treatment, and at 5, 30, and 60 Minutes Post-treatment
Description: The Injection Site Pain (during injection and post-injection) will be self-assessed by the subject using a 100 mm Visual Analog Scale (VAS). VAS is a 100 mm Visual Analog Scale with 0 meaning no pain and 100 meaning intolerable pain.
Time Frame: Immediately after treatment, and at 5, 30, and 60 minutes post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
Number analyzed (Participants) | 50 | 50
score on a scale
  Immediately after treatment | 34.7 (25.9) | 41.3 (25.8)
  5 minutes post-treatment | 3.5 (9.3) | 3.5 (8.9)
  30 minutes post-treatment | 1.3 (5.3) | 0.2 (1.4)
  60 minutes post-treatment | 0.4 (2.2) | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: across the duration of the study, approximately 12 weeks after last treatment (initial and touch up), up to 16 weeks
Arm/Group | RHA®4 - Cannula | RHA®4 - Needle
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 23/50 | 29/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHA®4 - Cannula (N=50) | RHA®4 - Needle (N=50)
Injection site induration (General disorders) | 13 (13) | 14 (14)
Injection site mass (General disorders) | 10 (13) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT04754646/Prot_001.pdf
  • Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT04754646/SAP_003.pdf